CLINICAL TRIAL: NCT02327819
Title: The Effect of Branched-chain Amino Acid (BCAA) on the Progression of Primary Liver Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 0440-14-TLV
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BCAA supplement (Active Comparator): Branched-chain amino acids supplement, 12 g/day
  Interventions: Dietary Supplement: Branched-chain amoni acids (BCAA)
- non-BCAA protein supplement (Sham Comparator): non-BCAA protein supplement
  Interventions: Dietary Supplement: non-BCAA protein supplement

INTERVENTIONS:
Dietary Supplement: Branched-chain amoni acids (BCAA)
  Arms: BCAA supplement
Dietary Supplement: non-BCAA protein supplement
  Arms: non-BCAA protein supplement

SUMMARY:
Supplementation of BCAA found to reduce the risk of developing liver cancer, but the affect of BCAA on existing liver cancer is unknown.

The participants (post curative intent surgery) will be supplemented with either BCAA/non-BCAA-enriched protein supplement. The intervantion will go on for 2 years or until a new liver tumor is found.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed primary liver cancer
* viral or Nonalcoholic Steatohepatitis Cirrhosis
* Cirrhosis rated Child-Pugh A
* liver cancer rated Barcelona Clinic Liver Cancer (BCLC) A

Exclusion Criteria:

* Age (over 65)
* liver condition rated Child-Pugh B/C
* GI/Absorption issues
* patients given a treatment before surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
time until a new liver tumor is found | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Unit, Sourasky Medical Center, Tel Aviv, Israel